CLINICAL TRIAL: NCT01459328
Title: Resource-Sparing Curative Treatment for Rectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Atomic Energy Agency (Other Government)
Collaborators: Centre Anti Cancer Hopital Frantz Fanon (Unknown); Hospital A.C. Camargo (Other); Credit Valley Hospital (Other); Instituto Nacional de Cancerologia, Columbia (Other Government); University Hospital Sestre Milosrdnice (Other); Minesterio de Cienca, Tecnologia y Medio Ambiente (Unknown); V.N. Cancer Center GKNM Hospital (Unknown); Tata Memorial Hospital (Other Government); Dr Cipto Mangunkusumo General Hospital (Other); National Cancer Center, Bratislava (Unknown); University of Cape Town (Other); Catholic University of the Sacred Heart (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E33034
Record Dates: First submitted 2011-10-10; First posted 2011-10-25 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Rectal Carcinoma
Keywords: rectal carcinoma; long course chemo-radiation; short course chemo-rdiation; Locally Advanced Rectal Carcinoma
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Conventional Long Course Chemo-Radiation (Active Comparator): Conventional long course chemo-radiation
  Interventions: Radiation: Radiotherapy
- Arm B: Short Course Radiation Followed by Chemotherapy (Experimental): Experimental short course radiation followed by chemotherapy.
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Short course radiotherapy: 25Gy in 5 daily fractions over 1 week Chemotherapy: - Bolus 5 Fluorouracil 450 mg/m2/day
  * Injected Leucovorin 20 mg/m2/day for 5 days
  Arms: Arm B: Short Course Radiation Followed by Chemotherapy
Radiation: Radiotherapy — Conventional long course chemo-radiation:
  * Radiation 50Gy in 25 daily fractions over 5 weeks
  * Bolus 5 Fluorouracil 350mg/m2/d for 5 days
  * Injected Leucovorin 20mg in both the first and last (5th) week of radiation
  * Oral Capecitabine (CAPE) 825mg/m2 b.i.d. during the entire radiotherapy course over 5 weeks.
  Arms: Arm A: Conventional Long Course Chemo-Radiation

SUMMARY:
This is a prospective, multicentre, randomized clinical trial comparing two different neo-adjuvant radiation-based strategies prior to intended surgery for locally advanced adenocarcinoma of the rectum.

This trial may establish the investigational therapy to be superior to, or at least not inferior to conventional treatment.

DETAILED DESCRIPTION:
This phase III randomised clinical trial compares the outcome of two different neo-adjuvant radiation based treatments for locally advanced rectal carcinoma. This encompasses patients at risk for a positive circumfrential resection margin (CRM+) on baseline assessment imaging and pateints identified as being with a T-descriptor T4 at baseline assessment.

The arms compared are as follows:

* The investigational arm: short chemo-radiation course(25Gy in 5 daily fractions over 1 week) +/- surgery.
* The conventional arm: protracted chemo-radiation course (50Gy in 25 daily fractions over 5 weeks combined with chemotherapy)+/- surgery.

The outcomes include four domains: overall survival, biological effect, quality of life and health-related economics.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Clinical (i.e. surgical determination) and/or diagnostic image findings consistent with c/uT4 or CRM+ (note that CRM+ must be established by MRI), primary rectal Adenocarcinoma (i.e. histology consistent with origin from rectal mucosa); these constitute LARC for the purpose of this protocol
* Treatment will be directed at the primary cancer, being clinically appropriate and given with an initial intent to cure the patient (this includes accepting up front that radiation and surgery are feasible; for surgery, this means that the patient has been determined fit for major surgery by an anaesthesiologist prior to the request for randomization)
* Performance status is sufficient to undertake the treatment in either arm (KPS>50%)
* Patient is accessible for required follow-up and data collection
* Radiation oncologist expects survival to exceed 6 months from date of diagnosis
* Patient provides informed consent

Exclusion Criteria:

* Recurrent rectal cancer
* Primary wholly in the sigmoid colon
* Considered to be arising in the anal canal
* Metastatic disease beyond the pelvis (by clinical assessment and/or diagnostic imaging)
* Contraindications to protocol RT or to protocol chemotherapy, such as one or more of the following:
* any prior RT to the pelvis; a solitary pelvic kidney within the intended radiation volume
* consideration by the most responsible radiation oncologist that the treatment volume is too large, or the amount of small bowel or other critical organs within the treatment volume is too much for safe treatment
* significantly abnormal laboratory tests such as impaired renal/liver function
* a haemoglobin that is < 8.0 (or 80, SI) and the patient is not transfused to exceed 8.0 (or 80, SI)
* on-going medications that are not compatible with protocol neo-adjuvant chemotherapy as described in this protocol
* Significant development issues (such as with age < 18 yr)
* Co-morbidity
* Psychiatric diagnosis
* Physical impairment
* Pregnancy or continuing breast-feeding, that precludes administration of protocol treatments, or that precludes data collection (such as likely to preclude follow-up visits or completing questionnaires)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2009-09; Primary Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | From commencement of radiation (day 1) to death or last follow-up up to 5 years.

SECONDARY OUTCOMES:
Biological Effect and Tumour Biology | Prior to surgical decision in weeks 13-15 and 4 weeks after surgery
  Maximum size of the tumor based on imaging and/or up to 3D measures reported by radiologists, comparing baseline and pre-surgical decision inverstigations
  If definitive surgery is conducted:
  * Proportion obtaining R0
  * Proportion undergoing TME
  * Status of the neurovascular and neural invasion(s)
  * Nodal ratio
  * Tumor sizes
  CEA results
Quality of Life | From date of randomization till the end of follow-up (5 years)
Health-related Economics | From date of randomization till the end of follow-up (5 years)
  Number of days in hospital
  Number of surgical procedures
  Number of days with stomas
  Protocol required therapies, as actually administered
  Adverse events that have significant cost implications (i.e. cost-drivers)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Rosenblatt, Principal Investigator — International Atomic Energy Agency
Locations (12):
- Centre Anti-Cancer, Hopital Franz Fanon, Blida, Algeria
- Hospital A.C. Camargo, Fundacao Antonio Prudente, São Paulo, Brazil
- Credit Valley Hospital, Mississauga, Ontario, Canada
- Instituto Nacional de Cancerologia, Minesterio de Salud, Bogota D.C., Colombia
- Department of Oncology and Nuclear Medicine, University Hospital Sestre Milosrdnice, Zagreb, Croatia
- Ministerio de Cienca, Tecnologia y Medio Ambiente (CITMA), La Habana, Cuba
- India (2):
  - Department of Radiation Oncology, V.N. Cancer Center, GKNM Hospital, Coimbatore
  - Department of Radiation Oncology, Tata Memorial Hospital, Mumbai
- Department of Radiotherapy, Dr. Cipto Mangunkusuma National General Hospital, University of Indonesia, Jakarta, Indonesia
- Instituto di Radiologia, Universita Cattolica del Sacro Cuore, Roma, Italy
- National Cancer Institute, Bratislava, Slovakia
- University of Cape Town, Cape Town, South Africa

REFERENCES:
- [Background] Bosset JF, Collette L, Calais G, Mineur L, Maingon P, Radosevic-Jelic L, Daban A, Bardet E, Beny A, Ollier JC; EORTC Radiotherapy Group Trial 22921. Chemotherapy with preoperative radiotherapy in rectal cancer. N Engl J Med. 2006 Sep 14;355(11):1114-23. doi: 10.1056/NEJMoa060829. PMID 16971718
- [Background] Kapiteijn E, Marijnen CA, Nagtegaal ID, Putter H, Steup WH, Wiggers T, Rutten HJ, Pahlman L, Glimelius B, van Krieken JH, Leer JW, van de Velde CJ; Dutch Colorectal Cancer Group. Preoperative radiotherapy combined with total mesorectal excision for resectable rectal cancer. N Engl J Med. 2001 Aug 30;345(9):638-46. doi: 10.1056/NEJMoa010580. PMID 11547717
- [Background] Radu C, Berglund A, Pahlman L, Glimelius B. Short-course preoperative radiotherapy with delayed surgery in rectal cancer - a retrospective study. Radiother Oncol. 2008 Jun;87(3):343-9. doi: 10.1016/j.radonc.2007.11.025. Epub 2008 Feb 21. PMID 18093674
- [Background] Braendengen M, Tveit KM, Berglund A, Birkemeyer E, Frykholm G, Pahlman L, Wiig JN, Bystrom P, Bujko K, Glimelius B. Randomized phase III study comparing preoperative radiotherapy with chemoradiotherapy in nonresectable rectal cancer. J Clin Oncol. 2008 Aug 1;26(22):3687-94. doi: 10.1200/JCO.2007.15.3858. PMID 18669453